CLINICAL TRIAL: NCT05242913
Title: A Randomized Double-blind, Placebo-controlled, Parallel Group Study to Evaluate the Effects of Resistant Potato Starch (SolnulTM) on Intestinal Flora
Brief Title: Effects of Resistant Potato Starch on the Gut Microbiota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MSP Starch Products Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: R10356
Record Dates: First submitted 2022-01-27; First posted 2022-02-16 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Microbiota
Keywords: Microbiota; Resistant Potato Starch; Bristol Stool Chart; Diarrhea; Constipation; Bloating; Abdominal Pain; Gas; Well-being
MeSH Terms: conditions — Diarrhea; Constipation; Abdominal Pain; Mucopolysaccharidosis IV

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Dose SolnulTM (Active Comparator): 7.0 g of Resistant Potato Starch administered daily for 4 weeks
  Interventions: Dietary Supplement: Resistant Potato Starch
- Low Dose SolnulTM (Active Comparator): 3.5 g of Resistant Potato Starch (plus 3.5 g digestible corn starch for 7.0 g total carbohydrate) administered daily for 4 weeks
  Interventions: Dietary Supplement: Resistant Potato Starch
- Placebo (Placebo Comparator): 7.0 g digestible corn starch administered daily for 4 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Resistant Potato Starch — Unmodified potato starch containing >60% resistant starch Type 2
  Other Names: Solnul; MSPrebiotic
  Arms: High Dose SolnulTM; Low Dose SolnulTM
Dietary Supplement: Placebo — Fully digestible corn starch
  Other Names: AmiocaTM
  Arms: Placebo

SUMMARY:
This was a randomized, double-blind, three-arm, parallel group clinical trial, which assessed the shifts that occur in microbial populations after four weeks of supplementation with resistant potato starch (SolnulTM) at two different dosages, in comparison to a placebo in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.0 and 34.9 kg/square meter (inclusive) that were generally healthy as determined by medical history and screening blood work.

Exclusion Criteria:

* Diagnosis of Irritable Bowel Syndrome (IBS), dyspepsia, significant gastrointestinal disorders, or other major diseases.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-01-06 (Actual)

PRIMARY OUTCOMES:
Changes in relative abundance (% of gut microbiome) of Bifidobacterium from stool between treatment groups | Four weeks
  Changes in relative abundance of Bifidobacterium after 4 weeks of consumption in High Dose, Low Dose, and placebo arms are compared.

SECONDARY OUTCOMES:
Changes in relative abundance (% of gut microbiome) of Bifidobacterium from stool between treatment groups | One week
  Changes in relative abundance of Bifidobacterium after 1 week of consumption in High Dose, Low Dose, and placebo arms are compared.
Changes in relative abundance (% of gut microbiome) of Bifidobacterium from stool within treatment groups | One week, four weeks
  Changes in relative abundance of Bifidobacterium between baseline and one or four week timepoints for High Dose, Low Dose, and Placebo arms.
Fecal SCFA (mmol/kg stool) changes from baseline | One week, four weeks
  Between and within group comparisons of SCFA levels in stool for High Dose, Low Dose, and Placebo arms
Changes from baseline in stool consistency using self-reported Bristol Stool Chart scores | One week, four weeks
  Changes in constipation and diarrhea frequency in High Dose, Low Dose, and Placebo arms.
Changes from baseline in gastrointestinal symptoms using the a modified Gastrointestinal Quality of Life Index scale | One week, four weeks
  Changes in bloating, belching, abdominal pain, gas, and overall well-being in High Dose, Low Dose, and Placebo arms.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Beir, MD, Principal Investigator — Nutrasource Pharmaceutical and Nutraceutical Services
Locations (1):
- Nutrasource Pharmaceutical and Nutraceutical Services, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bush JR, Alfa MJ. Consumption of resistant potato starch produces changes in gut microbiota that correlate with improvements in abnormal bowel symptoms: a secondary analysis of a clinical trial. BMC Nutr. 2024 Nov 27;10(1):152. doi: 10.1186/s40795-024-00962-7. PMID 39605008